CLINICAL TRIAL: NCT03002532
Title: Whole Brain Irradiation With Hippocampal Sparing for Brain Metastases From Breast Cancer: Neurocognitive Function and Prognosis Analysis
Brief Title: Hippocampal-sparing Whole Brain Radiotherapy for Brain Metastases From Breast Cancer
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Affiliated Hospital to Academy of Military Medical Sciences (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: ky-2016-9-37
Record Dates: First submitted 2016-12-20; First posted 2016-12-23 (Estimated); Last update posted 2016-12-23 (Estimated); Status verified 2016-12

CONDITIONS: Breast Cancer Metastatic; Brain Metastases
Keywords: Breast cancer; Brain metastasis; Whole brain radiotherapy; Hippocampal avoidance; Neurocognitive function; intracranial failure
MeSH Terms: conditions — Brain Neoplasms; Breast Neoplasms

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Whole-brain radiotherapy (WBRT) group (Active Comparator): Conventional whole-brain radiotherapy for brain metastases from breast cancer with dose of 37.5 Gy in 15 fractions.
  Interventions: Radiation: whole brain radiotherapy
- Hippocampal-sparing WBRT (HS-WBRT) group (Experimental): Hippocampal-sparing whole brain radiotherapy is performed using modern intensity-modulated radiotherapy (IMRT) technique to avoid conformally the hippocampal neural stem-cell structure during WBRT. Prescription dose is 37.5 Gy in 15 fractions.
  Interventions: Radiation: whole brain radiotherapy

INTERVENTIONS:
Radiation: whole brain radiotherapy

SUMMARY:
Based on evidence that radiation-induced damage to the hippocampus plays a considerable role in neurocognitive decline after cranial irradiation, hippocampal-sparing whole brain radiation therapy (HS-WBRT) has been proposed. This study will investigate the neurocognitive function and prognosis between HS-WBRT and conventional WBRT for the treatment of brain metastases from breast cancer.

ELIGIBILITY:
Inclusion Criteria:

* Female patients with advanced breast cancer who is confirmed historically.
* New developing brain metastases (BM) is confirmed by gadolinium contrast-enhanced magnetic resonance imaging (MRI), with or without clinical symptoms and pathology, and without a history of BM treatment.
* At least 2 BM lesions with the diameter of the largest lesion < 40 mm is eligible. And the distance from the border of a mass to the hippocampal margin should be more than 15 mm.
* The Eastern Cooperative Oncology Group (ECOG) is from 0 to 2, and the expected life expectancy is ≥3 months.

Exclusion Criteria:

* Concurrent chemoradiation.
* Patient who had received cranial irradiation previously.
* Patient who are enrolled in other clinical trial at the same time.
* Patient who has severe co-morbidity or infection.

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2015-08; Primary Completion 2017-08 (Estimated); Study Completion 2017-08 (Estimated)

PRIMARY OUTCOMES:
neurocognitive function | 1 years
  delayed recall using Hopkins Verbal Learning Test

SECONDARY OUTCOMES:
quality of life | 2 years
  Mini-Mental State Examination
patient-reported quality of life | 2 years
  Spitzer Quality of Life Index
time to intracranial progression | 2 years
overall survival after brain metastases | 2.5 years

CONTACTS AND LOCATIONS:
Overall Officials: Bing Sun, M.D., Principal Investigator — Affiliated Hospital of Academy of Military Medical Sciences
Locations (1):
- Affiliated Hospital of Academy of Military Medical Sciences, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Sun B, Huang Z, Wu S, Shen G, Cha L, Meng X, Ding L, Wang J, Song S. Incidence and relapse risk of intracranial metastases within the perihippocampal region in 314 patients with breast cancer. Radiother Oncol. 2016 Jan;118(1):181-6. doi: 10.1016/j.radonc.2015.11.010. Epub 2015 Dec 7. PMID 26674923
- [Result] Sun B, Huang Z, Wu S, Ding L, Shen G, Cha L, Wang J, Song S. Cystic brain metastasis is associated with poor prognosis in patients with advanced breast cancer. Oncotarget. 2016 Nov 8;7(45):74006-74014. doi: 10.18632/oncotarget.12176. PMID 27659537